CLINICAL TRIAL: NCT06691789
Title: Impact of Remote Social Support on Midwifery Students' Anxiety and Attitudes During Distance Education: a Randomized Study
Brief Title: Remote Social Support on Midwifery Students' Anxiety and Attitudes During Distance Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Elif Balkan, Research Assistant, Istinye University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: Istinye039
Record Dates: First submitted 2024-11-10; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2020-05

CONDITIONS: Anxiety
Keywords: anxiety; distance education; pandemics; COVID-19; social support
MeSH Terms: conditions — Anxiety Disorders; COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): This arm had intervention
  Interventions: Other: Social support
- Control (No Intervention): This arm had no intervention

INTERVENTIONS:
Other: Social support — This intervention includes a social support given to the students during COVID-19 pandemic
  Arms: Intervention

SUMMARY:
The aim of this CT is to evaluate the effects of distance social support program on anxiety and attitudes towards distance education with midwifery students during COVID-19. The main questions are:

1. Does online social support has an impact on attitudes towards distance education?
2. Does online social support decrease the anxiety levels of the students?

Participants will:

- Join an online social support program and meet the researchers and friends.

ELIGIBILITY:
Inclusion Criteria:

* Being 2nd or 3rd grade midwifery student
* voluntarily participating

Exclusion Criteria:

* not using smartphone

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Attitude Scale Towards Distance Education | From enrollment to the end of the study
  ASDE aims to assess the attitudes of the students towards distance education
Multidimensional Scale of Perceived Social Support | From enrollment to the end of the study
  MSPSS aims to assess the perceived social support.

SECONDARY OUTCOMES:
State and Trait Anxiety Scale | From enrollment to the end of the study
  STA-I aims to assess the anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not shared because of the ethical restrictions